CLINICAL TRIAL: NCT06532838
Title: Optimized Strategies for Acute Type A Aortic Dissection Complicated With MalPerfusion Syndrome (OPTIMIZE-MPS)
Brief Title: Optimized Strategies for Malperfusion Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Xijie Wu, Director, Head of Cardiovascular Surgery, Principal Investigator, Clinical Professor, Xiamen Cardiovascular Hospital, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (2024) YLK-26
Record Dates: First submitted 2024-07-26; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Aortic Dissection
Keywords: Malperfusion syndrome; Aortic dissection; Optimized strategies; Central repair; Endovascular reperfusion
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized treatment strategies (OTS group) (Experimental): Patients randomized to OTS group will be treated with optimized treatment strategies.
  Interventions: Procedure: Optimized treatment strategies
- Traditional treatment strategies (TTS group) (Active Comparator): Patients randomized to TTS group will be treated with traditional treatment strategies.
  Interventions: Procedure: Traditional treatment strategies

INTERVENTIONS:
Procedure: Optimized treatment strategies — The optimized strategies based on 6-hour threshold from symptom onset. For malperfused patients with symptom onset within 6 hours, central repair will be performed immediately. Additional stenting will be used in patients with persistent malperfusion. For malperfused patients with symptom onset beyond 6 hours, individualized delayed central repair according to the different types of MPS will be performed after organ function improved and the patient could tolerate central repair.
  Arms: Optimized treatment strategies (OTS group)
Procedure: Traditional treatment strategies — Immediate central repair will be performed for patients with coronary and cerebral malperfusion syndrome. However, for patients with mesenteric and lower extremity malperfusion syndrome, interventional therapy will be administered through fenestration and/or stenting to ﬁrst alleviate organ ischemia. Once the patients had a resolution of organ failure, corrective open aortic repair will be performed.
  Arms: Traditional treatment strategies (TTS group)

SUMMARY:
An investigator-initiated, randomized, multicenter, two-arm, open-label study of consecutive patients presenting with acute type A aortic dissection (ATAAD) and malperfusion syndrome (MPS).

Objectives: The present study aimed to investigate the difference in all-cause mortality after optimized treatment strategies (OTS) versus traditional treatment strategies (TTS) for ATAAD patients with MPS.

Background: The mortality of ATAAD with MPS is high. However, the management strategies of MPS patients still not to be confirmed. Compare with TTS, OTS as a strategy for ATAAD patients with MPS might have be beneficial results.

DETAILED DESCRIPTION:
A total of 236 subjects with ATAAD complicated with MPS who met inclusion criteria and do not have any exclusion criterion will be randomized to optimized treatment strategies (OTS) group and traditional treatment strategies (TTS) group.

1. Patients randomized to OTS group will be treated with optimized treatment strategies. The optimized strategies based on 6-hour threshold from symptom onset. For malperfused patients with symptom onset within 6 hours, central repair will be performed immediately. Additional stenting will be used in patients with persistent malperfusion. For malperfused patients with symptom onset beyond 6 hours, individualized delayed central repair according to the different types of MPS will be performed after organ function improved and the patient could tolerate central repair.
2. Patients randomized to TTS group will treated with traditional treatment strategies. Immediate central repair will performed for patients with coronary and cerebral malperfusion syndrome. However, for patients with mesenteric and lower extremity malperfusion syndrome, interventional therapy will be administered through fenestration and/or stenting to first alleviate organ ischemia. Once the patients had a resolution of organ failure, corrective open aortic repair will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures;
* Acute type A aortic dissection is confirmed by computed tomography angiography;
* The symptoms onset within 2 weeks;
* Patients are diagnosed with ATAAD, with a new diagnosis of malperfusion syndrome ,by meeting both of the following criteria:

  1. Radiographic findings reveal occlusion of the corresponding arteries (including either coronary artery, either carotid artery, celiac trunk, superior mesenteric artery or either iliac artery);
  2. Clinical features of end organ ischemia (altered consciousness, paralysis, melena, abdominal pain, tenderness to palpation, loss of sensory or motor function of the lower extremities) OR laboratory findings suggestive of end organ ischemia (elevated cardiac enzymes, lactate, myoglobin, or creatine kinase).

Exclusion Criteria:

* Age <18 yr and >80 yr;
* Unstable condition with cardiac tamponade or aortic rupture on admission;
* Multiple types of malperfusion syndrome on admission;
* Bloody stools or melena on admission;
* Bilaterally fixed dilated pupils, hemorrhagic infarction or herniation of brain on admission;
* Cardiopulmonary arrest and required continuous uninterrupted cardiopulmonary resuscitation on admission;
* Irreversible multiple organ failure on admission;
* Life expectancy < 1 year;
* Patients and (or) their families refused surgery;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Operative Mortality (OM) | 30-day
  Patients who died within 30 days

SECONDARY OUTCOMES:
Rate of composite of Major Adverse Events (MAE) | 30-day
  Number of participants with MAE which will include the composite rate of low cardiac output syndrome, new cerebrovascular accident, intestinal ischemia, lower limb necrosis, multiple organ failure according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Rate of composite of Major Adverse Pulmonary Events (MAPE) | 30-day
  Number of participants with MAPE which will include the composite rate of intubation >48 hours, pneumonia, reintubation, tracheostomy according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Rate of reintervention | 3 year
  The number of participants who will require reoperation for distal aorta
Mid-term survival | 3 year
  The secondary endpoint of the study is the evaluation of mid-term survival

CONTACTS AND LOCATIONS:
Locations (1):
- Xiamen Cardiovascular Hospital at Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided